CLINICAL TRIAL: NCT06480812
Title: The Role of a Synbiotic in Modulating Host Physiology Via the Gut Microbiome- A Pilot Randomised Controlled Dietary Intervention Study
Brief Title: The Role of Synbiotics in Modulating Host Physiology Via the Gut Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Simpson (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Organization: University of Nottingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FMHS 314-0623
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Intervention Model Description: Randomised Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic arm (Active Comparator): Synbiotic mixure (10g prebiotic fibre + 170ml kefir) will be randomly allocated to eligible participants in order to test specific effects of the synbiotic mixture on gut microbiome composition and metabolic markers.
  Interventions: Dietary Supplement: Synbiotic
- Control (Placebo Comparator): Individuals in the control arm will not be provided with the test supplement and asked to carry on with their usual diet and lifestyle.
  Interventions: Dietary Supplement: Synbiotic

INTERVENTIONS:
Dietary Supplement: Synbiotic — The proposed protocol will provide a simple but robust intervention study using a synbiotic (pre and probiotic combination) in order to improve our understanding of the mechanisms linking nutrition to health outcomes that are mediated by the gut microbiome.
  This pilot study will comprise a controlled randomised intervention in which participants will be grouped into the active synbiotic arm or the control arm. The ratios will be 10g of the prebiotic supplement and 170ml of kefir. Randomisation will control for equal distribution of age and biological sex; characteristics that may confound between group comparisons and will be assessed by analysis of baseline data.

SUMMARY:
The current study is a proof of concept mechanistic study that will utilise a combination of prebiotic and probiotic (synbiotic) supplements. The proposed study will improve our understanding of the molecular mechanisms linking nutrition to health outcomes that are mediated by the gut microbiome.

DETAILED DESCRIPTION:
The aim of this study is to generate high quality pilot data examining the role of a combination of pre and probiotic (synbiotic) supplementation in improving metabolic health (particularly systemic inflammation) and quality of life.

Specific Aim 1: To deliver a wealth of data, including effect sizes, on the physiological effects of synbiotic supplementation on the changes in the microbiome and metabolomic profile of an individual.

Specific Aim 2: To investigate potential mechanisms whereby the gut microbiome modulates crucial physiological parameters such as inflammatory markers and mental well-being measures.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participant eligibility includes those aged >18 years who have a body mass index (BMI) between 18.5 and 39.9 kg/m2
* Have a smart phone in order to download apps on phone

Exclusion Criteria:

* Have any gastrointestinal condition or food intolerance which could impact ability to comply with the intervention (e.g. IBS, malabsorptive conditions such as IBD, coeliac)
* Have lactose intolerance
* Have diabetes mellitus or any condition with an inflammatory component such as asthma, psoriasis, arthritis etc.
* Are currently taking fibre or probiotic supplements
* Are taking any prescribed medication
* Are currently following or anticipated to commence a specialised commercially available weight loss diet and/or program
* Are pregnant or breast feeding
* Currently have a diagnosed psychiatric illness
* History or current neurological condition (e.g. epilepsy)
* Have taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Change in systemic inflammatory profile | 6 weeks
  Change in circulating markers of systemic inflammation in serum samples collected pre and post the 6-week intervention period.

SECONDARY OUTCOMES:
Change in gut microbiome profile | 6 weeks
  Change in gut microbiome profile, assessed using 16s RNA sequencing analysis of faecal samples provided pre and post the 6-week intervention period
Changes in short chain fatty acids (SCFAs) | 6 weeks
  Change in serum SCFAs measured by mass spectrometry pre and post the 4-week intervention period
Mental Wellbeing as measured by validated questionnaires | 6 weeks
  The Hospital Anxiety and Depression Survey (HADS) was used to assess subjective measures of anxiety and depression. The scores for each subscale (HADS-Anxiety (A) and HADS-Depression (D)) range from 0 to 21. The cut-off scores range from:
  0-7: Normal (no significant symptoms) 8-10: Borderline or mild symptoms 11-21: Clinically significant anxiety or depression
Changes in skin microbiome profile | 6 weeks
  Change in skin microbiome profile, assessed using 16s RNA sequencing analysis of faecal samples provided pre and post the 6-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Vijay, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data arising from the current study will be fully anonymised and used for publication purposes

REFERENCES:
- [Derived] Vijay A, Simpson L, Tooley M, Turley S, Kouraki A, Kelly A, Menni C, Armstrong J, Jones S, Valdes AM. The anti-inflammatory effects of three different dietary supplement interventions. J Transl Med. 2025 Oct 16;23(1):1081. doi: 10.1186/s12967-025-07167-x. PMID 41094562